CLINICAL TRIAL: NCT04564963
Title: The Effect of Intermittent Cryotherapy Exposure (ICE) on Patients' Quality of Recovery After Surgery: A Vanguard Randomized Control Trial
Brief Title: The Effect of Intermittent Cryotherapy Exposure on Patients' Quality of Recovery After Surgery
Acronym: ICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Paul Karanicolas, Scientist and Associate Professor, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO Project ID 2021
Record Dates: First submitted 2020-09-08; First posted 2020-09-25 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain
Keywords: Cryotherapy; Cold therapy; Pain management
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Multi-centre, pragmatic, open label, two-arm parallel-group Vanguard feasibility randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy (Experimental): Cold therapy
  Interventions: Other: Cryotherapy
- No cryotherapy (No Intervention): Standard practices for pain management

INTERVENTIONS:
Other: Cryotherapy — Application of cryotherapy (e.g. ice in resealable zipper storage bags, gel packs, ice packs) over largest closed incision in the post-operative period every 4 hours, at minimum, for up to 72 hours (while participant is awake and admitted to hospital). The cryotherapy should not be placed in direct contact with skin.
  Arms: Cryotherapy

SUMMARY:
"Cryotherapy", or cold therapy, can include the use of gel packs, ice bags, ice baths, whole body chambers, and cold aerosol sprays. It is a popular non-drug treatment that can be used after a surgical operation, along with medication such as narcotics and anti-inflammatories for pain management. The application of ice packs on areas of injury has been used for many decades, as they can decrease both inflammation and pain. Other possible benefits include reduced blood flow, swelling, and tissue damage as well as muscle spasms. While there is some evidence to suggest that the use of ice packs is beneficial, this has not yet been implemented into practice, nor do any guidelines recommend the use of ice packs for pain management in surgical patients. In this trial, adult patients undergoing scheduled thoracoabdominal or groin surgery will be randomly assigned to apply ice packs over the largest closed surgical incision every 4 hours, at minimum, for 72 hours (while the patient is awake), along with standard of care, or to receive standard of care only. This trial will be conducted under the IMPACTS (Innovative, Multicentre, Patient-centred Approach to Clinical Trials in Surgery) program umbrella and will follow IMPACTS methodology. For the Vanguard trial, the aim is to determine the feasibility of conducting a definitive trial. Future outcomes of interest are quality of patient recovery, pain, length of hospital stay and medication use.

DETAILED DESCRIPTION:
Background/rationale: To date, there is some evidence to suggest a benefit of cryotherapy application over closed post-operative incisions, however, this has not yet been implemented into practice. Furthermore, there are no clinical practice guidelines that recommend the application of cryotherapy for adjuvant pain management. Relevant randomized controlled trials (RCTs) in abdominal surgery demonstrate a possible advantage of cryotherapy application, when compared to no cryotherapy application. However, those RCTs were small and were restricted to gynecology procedures or emergent procedures. Therefore, the investigators aim to address this knowledge gap by assessing the benefit of applying cryotherapy post-operatively (along with standard of care approaches), compared to no cryotherapy, (i.e., standard of care, only) over closed incisions, across broad surgical specialties and procedures, to improve the quality of patient recovery in adult patients.

Objectives: Before embarking on a definitive RCT, this pilot trial has five specific feasibility objectives:

1. To assess the investigators' ability to accrue patients using the IMPACTS Program design platform at multiple institutions, over the course of one year.
2. To assess the investigators' ability to adaptively randomize patients and deliver the randomized assignment using the IMPACTS Program design platform, over the course of one year.
3. To assess the investigators' ability to collect complete data directly from participants (patients and clinicians) on: narcotics use and surgical site infections over the course of one year.
4. To examine the investigators' ability to carry out data linkages using the IMPACTS Program design platform over the course of one year.
5. To estimate the change in quality of recovery to inform the sample size calculation for the definitive trial.

Study design: This is a multicentre, pragmatic, open label, two-arm parallel-group Vanguard feasibility randomized controlled trial. Patients will be randomized to cryotherapy application or no cryotherapy application. If feasibility is demonstrated during the pilot trial, the investigators will plan to conduct a definitive trial. If there are only minimal changes to the protocol, the investigators will include data from the pilot phase into the definitive trial analysis (i.e. a Vanguard design).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Scheduled for an elective surgery requiring a thoracic, abdominal or groin incision
* Scheduled to remain in hospital for at least one night, post-operatively

Exclusion Criteria:

* Anticipated to require intubation overnight post-operatively
* Raynaud's phenomenon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-08-21 (Actual)

PRIMARY OUTCOMES:
Assessment of accrual (one year) | 1 year
  Average number of patients enrolled per month across the 3 sites for the trial: feasible if 10 or more
Proportion of participants who received the allocated intervention, across all sites | 1 year
  Feasible if >90% of patients receive correct intervention
Proportion of complete data collection for patient-reported outcome surveys, across all sites | 1 year
  Feasible if >80% of data is collected
Proportion of successful data linkage of patient-reported outcome data with Institute of Clinical Evaluative Sciences and National Surgical Quality Improvement Program dataset(s), across all sites | 1 year
  Feasible if linkage is possible in >90% of patients
Estimation of Quality of Recovery (QoR) in patients treated with cryotherapy vs. no cryotherapy | 1 year
  Quality of patient recovery will be measured using the QoR-15 score at post-operative day 1 (POD1). The QoR-15 score ranges from 0-150 (the higher the score, the better the recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Karanicolas, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- Canada (3):
  - North York General Hospital, North York, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No